CLINICAL TRIAL: NCT00434187
Title: An Ascending Multiple Dose Study of the Safety, Tolerability and Pharmacokinetics of ERB-041 Administered Orally to Healthy, Female Japanese Subjects
Brief Title: Study to Evaluate Multiple Doses of ERB-041 in Healthy, Female Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3142A2-115
Record Dates: First submitted 2007-02-09; First posted 2007-02-13 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Healthy
Keywords: healthy
MeSH Terms: interventions — ERB 041

INTERVENTIONS:
Drug: ERB-041

SUMMARY:
The primary objective is evaluate the safety, tolerability, and pharmacokinetics of multiple doses of ERB-041, an investigational drug, in healthy, female Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by the investigator on the basis of medical history and screening evaluations.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24
Dates: Start 2006-08; Study Completion 2006-10

PRIMARY OUTCOMES:
safety, pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Kan-nondai, Tsukuba-shi, Ibaraki, Japan